CLINICAL TRIAL: NCT00576888
Title: International Registry for Vascular Anomalies Associated With Coagulopathy
Brief Title: Registry for Vascular Anomalies Associated With Coagulopathy
Acronym: VAC
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Beth A Drolet, MD, Professor of Dermatology and Pediatrics, Medical College of Wisconsin
Other Study IDs: CHW07/226
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Multifocal Lymphangioendotheliomatosis With Thrombocytopenia; Cutaneovisceral Angiomatosis With Thrombocytopenia; Vascular Anomaly With Thrombocytopenia; Hemangiomas
Keywords: Multifocal lymphangioendoltheliomatosis with thrombocytopenia; Cutaneovisceral angiomatosis with thrombocytopenia; Thrombocytopenia; Hemangiomas; Hemangiomatosis; Lymphatic malformation; Kasabach-Merritt; Blue-rubber bleb nevus; Angiomatosis
MeSH Terms: conditions — Hemangioma; Thrombocytopenia; Lymphatic Abnormalities; Blue rubber bleb nevus syndrome; Angiomatosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Buccal swab, tissue biopsy if available
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vascular Anomaly with Coagulopathy: All patients diagnosed with Multifocal lymphangioendotheliomatosis with thrombocytopenia (MLT) or with a vascular anomaly with coagulopathy
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention - observational only

SUMMARY:
PURPOSE The purpose of this study is to learn more about multifocal lymphangioendotheliomatosis with thrombocytopenia (MLT). MLT is a rare vascular disorder characterized by multiple congenital skin and visceral lesions, profound thrombocytopenia, and gastrointestinal bleeding. The skin lesions may appear red, brown or blue, often misdiagnosed as hemangiomas. The gastrointestinal tract, liver, and lungs are the most common internal organs involved. The severe thrombocytopenia (low platelets) is believed to be the result of platelet trapping within the skin and visceral vascular lesions. Severe and chronic gastrointestinal bleeding is common during infancy and early childhood. Although a relatively newly described entity, MLT was likely previously reported as hemangiomas, blue rubber bleb nevus syndrome, diffuse hemangiomatosis, Kasabach-Merritt phenomenon, and hereditary hemorrhagic telangiectasia. The term cutaneovisceral angiomatosis with thrombocytopenia is also a term used for this same disease. This study is a longitudinal cohort study of MLT to collect detailed clinical data on the distribution of disease, disease severity, and complications. This data will be used to create diagnostic criteria and an evaluation protocol for infants with this disease

DETAILED DESCRIPTION:
After informed consent is obtained a detailed question will be mailed to participating patients and families. This questionnaire will also be available electronically through an educational website. Data collected will include photographs of skin lesions, video images of gastrointestinal lesions, demographic data, clinical information, therapeutic interventions, glass slides of tissue biopsies, and collection of DNA. Enrollment will be patient family driven and modeled after several successful registries of rare diseases.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a vascular anomaly with coagulopathy

Exclusion Criteria:

* Subjects without a vascular anomaly with coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with Multifocal lymphangioendotheliomatosis with thrombocytopenia (MLT) or with a vascular anomaly with coagulopathy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2018-12 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with genetic mutations, copy number variations and/or expression analysis | After DNA collected and batches are sent for analysis
  Expand knowledge on consensus diagnostic criteria, atypical presentations and long term outcomes of patients with vascular anomalies

CONTACTS AND LOCATIONS:
Overall Officials: Beth Drolet, MD, Principal Investigator — Medical College of Wisconsin; Ulrich Broeckel, MD, Principal Investigator — Medical College of Wisconsin; Howard Jacob, PhD, Principal Investigator — Medical College of Wisconsin; Michael Kelly, MD, PhD, Principal Investigator — Medical College of Wisconsin; Richard Noel, MD, PhD, Principal Investigator — Medical College of Wisconsin; Paula North, MD, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States